CLINICAL TRIAL: NCT00813618
Title: Phase I Study of MEDI 507 in the Treatment of Pediatric Patients With at Least Grade II Acute Graft-Versus-Host Disease (GvHD)
Brief Title: Study of MEDI 507 in the Treatment of Pediatric Patients
Acronym: Pediatric GvHD
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: MedImmune LLC (Industry)
Responsible Party: Christine A. Dingivan, MD, Medimmune LLC
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MI-CP049
Record Dates: First submitted 2008-12-19; First posted 2008-12-23 (Estimated); Last update posted 2008-12-23 (Estimated); Status verified 2008-12

CONDITIONS: Graft Versus Host Disease
Keywords: Acute GvHD of at least Grade II severity
MeSH Terms: conditions — Graft vs Host Disease | interventions — siplizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental): MEDI-507
  Interventions: Drug: MEDI-507
- 2 (Experimental): MEDI-507
  Interventions: Drug: MEDI-507
- 3 (Experimental): MEDI-507
  Interventions: Drug: MEDI-507

INTERVENTIONS:
Drug: MEDI-507 — 0.012 mg/kg given intravenously on Study Days 0, 3, 6 and 9
  Arms: 1
Drug: MEDI-507 — 0.04 mg/kg given intravenously on Study Days 0, 3, 6 and 9
  Arms: 2
Drug: MEDI-507 — 0.12 mg/kg given intravenously on Study Days 0, 3, 6 and 9
  Arms: 3

SUMMARY:
To assess the safety of escalating dose levels of MEDI-507 in pediatric stem cell and bone marrow allograft recipients who have at least Grade II GvHD.

DETAILED DESCRIPTION:
This is a Phase I, open-label dose escalation trial of MEDI-507 in pediatric SCT and BMT recipients with at least Grade II acute GvHD. All patients will receive steroid therapy and MEDI-507 for treatment of GvHD

ELIGIBILITY:
Inclusion Criteria:

* Allogeneic BMT or SCT recipients
* Acute GvHD of at least Grade II severity
* Age 2 to 17 years
* Evidence of engraftment (ANC over 500 cells/mm3 on two consecutive days within seven days before study entry)
* Receipt of GvHD prophylaxis regimen including methotrexate, tacrolimus or cyclosporine
* Receipt of at least 2 mg/kg of methylprednisolone (or equivalent corticosteroid) between eight and 24 hours prior to the first MEDI-507 dose for GvHD treatment
* Both males and females are eligible, but sexually active females at risk of pregnancy of childbearing potential must agree to use an effective method of avoiding pregnancy (which includes oral or implanted contraceptives, IUD, female condom, diaphragm with spermicide, cervical cap, abstinence, use of a condom by the sexual partner or sterile sexual partner) beginning 30 days before the first study infusion and continuing through 60 days after the final study infusion.

Exclusion Criteria:

* Treatment of acute GvHD with methylprednisolone (or equivalent corticosteroid) at a total dose exceeding 14 mg/kg (or equivalent) over a seven day period (for example, 2 mg/kg/day for seven days)
* Previous receipt of MEDI 507
* Previous treatment with any anti-T cell monoclonal antibodies, such as OKT3, daclizumab (Zenapax), or basiliximab (Simulect)
* Treatment with anti-thymocyte globulin (ATG, ATGAM or others) within 14 days
* More than one allogeneic bone marrow or hematopoietic stem cell allograft
* Use of other investigational agents within 30 days (this does not include the use of licensed agents for indications not listed in the package insert) or current participation in a research protocol in which an investigational agent was administered
* Any of the following clinical settings or diagnoses:
* documented or presumed significant active infection
* pregnancy or nursing mother
* evidence of infection with HIV-1, hepatitis B or C virus
* hemodialysis or chronic peritoneal dialysis
* use of a ventilator
* chronic GvHD
* active veno-occlusive disease of the liver
* moribund patient

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 10 (Actual)
Dates: Start 1999-09; Primary Completion 2004-06 (Actual); Study Completion 2004-08 (Actual)

PRIMARY OUTCOMES:
Safety assessment of escalating dose levels of MEDI-507 in pediatric stell scell (SCT) and bone marrow (BMT) allograft recipients who have at least Grade II Graft-versus-Host Disease (GvHD). | Through Study Day 44

SECONDARY OUTCOMES:
Evaluate the serum concentrations and pharmacokinetics (PK) of MEDI 507 and pharmacodynamic effects of MEDI-507 on the absolute lymphocyte count and dynamics of lymphocyte phenotypes. | Through Study Day 364

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - Children's Hospital, Birmingham, Alabama
  - Children's Hospital of Orange County, Orange, California
  - Children's Memorial Hospital, Chicago, Illinois
  - Univ. of Michigan Medical Center, Ann Arbor, Michigan
  - Hackensack U. Medical Center, Hackensack, New Jersey
  - The Children's Hosp. of Phila., Abramson Ped. Research Center, Philadelphia, Pennsylvania